CLINICAL TRIAL: NCT01750320
Title: Koning Breast CT-guided Biopsy Phase I Trial
Brief Title: Koning Breast Computed Tomography Guided Biopsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Koning Corporation (Industry)
Collaborators: Elizabeth Wende Breast Care, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KBCT-004; W81XWH-09-1-0441 (Other Grant/Funding Number: Department of Defense (DOD) Telemedicine and Advanced Technology Research Center (TATRC))
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Breast CT; Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Koning Breast CT - guided Biopsy (Experimental)
  Interventions: Device: Koning Breast CT-guided Biopsy

INTERVENTIONS:
Device: Koning Breast CT-guided Biopsy — The breast will be positioned and stabilized in the grid/compression device. Four KBCT scans will be taken to guide the vacuum-assisted biopsy procedure.

SUMMARY:
The primary aim of this study is to show that the accuracy of Koning Breast CT-guided biopsy is at least equivalent to that of stereotactic-guided biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 35 years of age of any ethnicity
* Lesion seen on mammography
* Diagnostic report read as BI-RADS 4 or 5
* Will undergo biopsy no later than four weeks from date of mammogram
* Is able to undergo informed consent

Exclusion Criteria:

* Pregnancy
* Lactation
* Subjects with breast implants
* Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pacemaker.
* Subjects who are unable to tolerate study constraints.
* Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkins disease
* Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The accuracy of Koning breast CT-guided biopsy | about 1 year
  The goal of this study is to evaluate the concordance of Koning Breast CT-guided Biopsy (KBCT-GBx) results to diagnostic work-up imaging (at least mammographic) and KBCT imaging and to verify that the localization and guidance accuracy of KBCT-GBx is at least equivalent to stereotactic-guided biopsy to validate the localization and guidance accuracy of KBCT-GBx.

CONTACTS AND LOCATIONS:
Locations (1):
- Elizabeth Wende Breast Care, Rochester, New York, United States